CLINICAL TRIAL: NCT07252570
Title: Portal Vein Stenting for Malignant Obstruction: Feasibility, Safety, and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Radio01
Record Dates: First submitted 2025-09-08; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Neoplasms; Pancreatic Neoplasm; Portal Hypertension; Portal Vein Thrombosis
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with malignant portal vein stenosis/occlusion treated by stent
  Interventions: Device: Transhepatic portal vein stent implantation

INTERVENTIONS:
Device: Transhepatic portal vein stent implantation — The intervention consisted of percutaneous transhepatic implantation of a self-expanding metallic stent in the portal vein to treat malignant symptomatic portal vein stenosis or occlusion. Patients were selected on the basis of clinical complications related to portal hypertension, such as refractory ascites or gastrointestinal bleeding. The procedure aimed to restore portal vein patency and reduce symptoms. Stents of different lengths (40 mm, 60 mm, or 80 mm) were deployed depending on the anatomical extent of the obstruction. All procedures were performed by interventional radiologists under image guidance. Patients were subsequently followed for technical success, stent patency, clinical efficacy, and procedure-related safety.

SUMMARY:
Introduction:

Pre-hepatic portal hypertension of malignant origin can lead to severe complications such as refractory ascites or gastrointestinal bleeding, significantly impairing patients' quality of life. Available therapeutic options are mainly symptomatic and do not address the venous obstruction. Portal vein stenting represents a minimally invasive alternative, which remains poorly studied in this setting. The aim of our study was to evaluate portal stent patency, as well as clinical efficacy and safety, in patients with symptomatic malignant stenosis or occlusion of the portal system. Methods: The team conducted a retrospective cohort study including 63 consecutive patients treated between April 2004 and March 2024 at CHU l'Archet and CAL Nice for symptomatic malignant stenosis or occlusion of the portal system. All patients underwent percutaneous transhepatic portal vein stenting with uncovered self-expandable metallic stents. The primary endpoint was stent patency, defined as the interval between implantation and the occurrence of an occlusion confirmed by imaging or end of follow-up. Secondary endpoints included technical success, clinical success (improvement of portal hypertension signs), and the occurrence of adverse events, graded according to the 2017 SIR classification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of symptoms related to portal hypertension (e.g., refractory ascites, gastrointestinal bleeding).
* Imaging evidence of stenosis or obstruction of the portal venous system (main portal vein, superior and/or inferior mesenteric vein, spleno-mesenteric confluence, and/or splenic vein).

Exclusion Criteria:

* Obstruction or stenosis secondary to a malignant/neoplastic process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of consecutive adult patients referred to the Interventional Radiology Department of Nice University Hospital (CHU l'Archet, France) between April 2004 and March 2024. All patients presented with symptomatic portal hypertension related to malignant portal venous stenosis or occlusion and were treated with percutaneous transhepatic portal vein stenting. Patients were identified retrospectively from institutional medical records.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2004-04-08 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Portal vein stent patency. | From stent placement until death or loss to follow-up to 110 months.
  Stent patency was assessed using cross-sectional imaging and/or Doppler ultrasound.

SECONDARY OUTCOMES:
Clinical efficacy (physiological parameter) of portal vein stenting | From stent placement until death or loss to follow-up to 110 months.
  Assessment was performed retrospectively using medical records, imaging studies, and follow-up endoscopy when available.
Safety of portal vein stenting. | From procedure date until last follow-up to 110 months and graded according to SIR 2017 classification
  Procedure-related adverse events were retrospectively collected from medical records and classified according to the Society of Interventional Radiology (SIR) complication grading system. Safety was assessed by recording the occurrence, type, and severity of adverse events following stent placement.
Technical success | From stent placement start to completion portography (1 hour).
  Successful stent implantation was defined as placement at the intended anatomical site with confirmed patency on completion portography.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, Alpes Maritimes, France